CLINICAL TRIAL: NCT00214240
Title: The Impact of Cytogam® on Time to Viral Load Reduction in Kidney or Kidney/Pancreas Transplant Recipients With Clinical CMV Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1999-492
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Cytomegalovirus
MeSH Terms: interventions — cytomegalovirus-specific hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cytogam in addition to standard of care (IV ganciclovir therapy)
  Interventions: Drug: CMV Immune globulin
- 2 (No Intervention): Receive standard of care therapy (IV ganciclovir)

INTERVENTIONS:
Drug: CMV Immune globulin — CMV IvIg 150mg/kg x 6 doses
  Arms: 1

SUMMARY:
This pilot study is to assess whether using CytoGam® in combination with ganciclovir is more effective in reducing the CMV viral load over time, as compared to standard treatment with IV ganciclovir only. Serial blood samples are drawn to measure the amount of CMV viral load weekly, while the subject is receiving treatment with ganciclovir, or ganciclovir + CytoGam®. Additional CMV viral load blood sampling (CMV DNA capture qualitative testing only) will occur weekly thereafter until the subject is 8 weeks from the time of CMV diagnosis or until the CMV infection is no longer detectable, whichever is longer duration.

ELIGIBILITY:
Inclusion Criteria:

* Renal or renal/pancreas transplant patients who are diagnosed with symptomatic CMV infection
* receiving no more than 48 hrs of therapy prior to study enrollment

Exclusion Criteria:

* serum creatinine <2.2 at the time of enrollment
* no prior use of CMV IgG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2000-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
CMV viral load | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John Pirsch, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States